CLINICAL TRIAL: NCT01157754
Title: Cycle Planning With OCP in GnRH Antagonists Cycles Versus Long Protocol in Good Prognosis IVF Patients
Brief Title: Oral Contraceptive Pill and GnRH Antagonist Versus Long Protocol in IVF Patients
Acronym: Larganta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IVI Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAD-GV-05-2009-01
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Infertility
Keywords: Infertility patients requiring IVF; good prognosis
MeSH Terms: conditions — Infertility | interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OCP+GnRH antagonist (Experimental): Microgynon 14 to 21 tablets starting COH on day 5 post pill, rFSH + GnRH antagonist
  Interventions: Drug: levonorgestrel and ethynilestradiol
- long GnRH agonist (Active Comparator): daily triptorelin starting day 21st of previous cycle
  Interventions: Drug: levonorgestrel and ethynilestradiol

INTERVENTIONS:
Drug: levonorgestrel and ethynilestradiol

SUMMARY:
Recent controversy has arisen regarding the use of the pill for cycle planning in GnRH antagonist IVF cycles. The investigators performed this study to compare such a protocol with the gold-standard still today, which is the long-agonist protocol with no previous use of the pill.

ELIGIBILITY:
Inclusion Criteria:

* 1st or 2nd IVF cycle
* BMI <30 kg/m2
* regular menstrual cycles
* basal FSH <10 IU and E2 <60 pg/ml

Exclusion Criteria:

* Polycystic ovaries
* endometriosis
* previous ovarian surgery
* previous low ovarian response

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
implantation rate | 2 weeks after the embryo transfer

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Valenciano de Infertilidad, Madrid, Madrid, Spain